CLINICAL TRIAL: NCT01657890
Title: A Phase 1, Open Label, Parallel Group, Single Dose Study to Evaluate the Pharmacokinetics of Isavuconazole in Healthy Non-Elderly and Elderly Male and Female Subjects
Brief Title: Study of the Pharmacokinetics of Isavuconazole in Healthy Non-Elderly and Elderly Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 9766-CL-0041
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Pharmacokinetics of Isavuconazole; Healthy Volunteers; Safety and Tolerability in Elderly
Keywords: isavuconazole; BAL8557
MeSH Terms: interventions — isavuconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: Isavuconazole in healthy non-elderly male subjects (Experimental): age 18 to 45 years
  Interventions: Drug: isavuconazole
- Arm 2: Isavuconazole in healthy non-elderly female subjects (Experimental): age 18 to 45 years
  Interventions: Drug: isavuconazole
- Arm 3: Isavuconazole in healthy elderly male subjects (Experimental): age 65 years and older
  Interventions: Drug: isavuconazole
- Arm 4: Isavuconazole in healthy elderly female subjects (Experimental): age 65 years and older
  Interventions: Drug: isavuconazole

INTERVENTIONS:
Drug: isavuconazole — oral
  Other Names: BAL8557

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of isavuconazole in healthy non-elderly and elderly male and female subjects.

DETAILED DESCRIPTION:
All subjects receive a single dose of isavuconazole on Day 1 under fasting conditions. Subjects are confined to study center from Day -1 until Day 4 when they are discharged. Subjects return for outpatient visits on Days 6, 8, 11, 13 and 15.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are healthy, non-elderly males and females between 18 and 45 years and healthy, elderly males and females 65 years of age and older
* The subject has a body weight of at least 45 kg and has a body mass index (BMI) of 18 to 32 kg/m2, inclusive
* The estimated (calculated) creatinine clearance must be within the age-appropriate normal range, if abnormal, the abnormality is not clinically significant, as determined by the Investigator
* Results for aspartate aminotransferase (AST) and alanine aminotransferase (ALT), and total bilirubin must be within the normal range
* The Female subject agrees to sexual abstinence, or is surgically sterile, postmenopausal (defined as at least 2 years at Screening without menses), or using a medically acceptable double barrier method (e.g. spermicide and diaphragm, or spermicide and condom) to prevent pregnancy and agree to continue using this method from Screening until 3 weeks after the follow-up visit at the end of the study; and is not lactating or pregnant as documented by negative pregnancy tests at Screening and Day -1
* The Male subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy and agrees to continue using this method from Screening until 3 weeks after the follow-up visit at the end of the study

Exclusion Criteria:

* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes)
* The subject has a positive result for hepatitis C antibodies, hepatitis B surface antigen at Screening or is known to be positive for human immunodeficiency virus (HIV)
* The subject has a known or suspected allergy to any of the components of the trial products including the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods (as judged by the investigator), or a history of severe anaphylactic reactions
* The subject is a smoker (any use of tobacco or nicotine containing products) within 6 months prior to Screening
* The subject, if non-elderly, has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Day -1, or over-the-counter medications within 1 week prior to Day -1, with the exception of acetaminophen up to 2 g/day
* The subject, if elderly, has not been on stable concomitant medications (minor necessary dosing changes are acceptable) for at least 4 weeks prior to study drug administration or is taking any medication that would interfere with the evaluation of isavuconazole in this study (CYP3A4 inducer or inhibitor)
* The subject has a recent history (within the last 2 years) of drug or alcohol abuse, as defined by the investigator, or a positive drug and/or alcohol screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) variables for isavuconazole (in plasma): AUCinf, AUClast, and Cmax | Day 1: Pre-dose, 0.5, 1, 1.5, 2, 3, 4 ,6, 8,10, 12, 16, 20, 24, 36, 48, 72, 120, 168, 240, 288, 336 hours post-dose on Day 1
  Area under the concentration-time curve from time of dosing to infinity (AUCinf), Area under the concentration-time curve from time of dosing to the last quantifiable concentration (AUClast) and Maximum concentration (Cmax)

SECONDARY OUTCOMES:
PK variables for isavuconazole (in plasma): Vz/F, CL/F, t1/2, tmax | Day 1: Pre-dose, 0.5, 1,1.5, 2, 3, 4, 6, 8,10, 12, 16, 20, 24 ,36, 48, 72, 120, 168, 240, 288, 336 hours post-dose on Day 1
  Apparent volume of distribution (Vz/F), Apparent body clearance after oral dosing (CL/F), Apparent terminal elimination half-life (t ½), Time to attain maximum concentration (tmax)
Safety assessed by recording adverse events, laboratory assessments, physical examinations, vital signs, electrocardiograms (ECGs) | Day 1-15

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Parexel International, Glendale, California, United States

REFERENCES:
- [Derived] Desai AV, Han D, Kowalski DL, Lademacher C, Pearlman H, Yamazaki T. No Dose Adjustment for Isavuconazole Based on Age or Sex. Antimicrob Agents Chemother. 2019 May 24;63(6):e02629-18. doi: 10.1128/AAC.02629-18. Print 2019 Jun. PMID 30962330